CLINICAL TRIAL: NCT06679530
Title: Music During Allogeneic Stem Cell Transplant Hospitalization: A Pilot Trial
Brief Title: Music During Allogeneic Stem Cell Transplant Hospitalization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-0862.cc
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Cell Transplantation (HCT)

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups including mindful music listening or standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention (Experimental)
  Interventions: Other: Mindful Music Listening (MML)
- Control (No Intervention)

INTERVENTIONS:
Other: Mindful Music Listening (MML) — Self-guided mindful music listening intervention comprised of 1-hour daily music listening during inpatient hospitalization.
  Arms: Music Intervention

SUMMARY:
The goal of this trial is to develop an Independent Music Listening tool for stem cell transplant patients that have prolonged hospitalizations. The main questions it aims to answer are:

[primary hypothesis or outcome measure 1]? [primary hypothesis or outcome measure 2]?

Participants will use a self-guided music listening intervention of 1-hour daily music listening during their inpatient hsopitalization and delivered via web-based platform.

DETAILED DESCRIPTION:
To address this clinical and research need in the current project, the primary aim is to (1) assess the feasibility, acceptability, and appropriateness of a self-guided music listening intervention (i.e. Independent Music Listening or "IML") comprised of 1-hour daily music listening during the inpatient hospitalization (e.g., 3-4 weeks) and delivered via web-based platform/smart phone app (e.g., Spotify or Apple music) among 35 HCT patients. Participants will be randomized to IML (n=23) or usual care control group (n=12). The secondary aims are to (2a) explore whether the IML program is associated with improvements on psychosocial self-report measures of patient quality of life, distress, and mindfulness and (2b) whether preliminary psychosocial effects of the IML program are different from a control group of patients completing usual care. In an exploratory aim, the PI will gather qualitative data on patient perceptions and reactions to daily music listening via a daily music diary and post-intervention open-ended questions. Data produced from the current study will help inform development of future interventions to improve quality of life in HCT patients that are based in arts in medicine or creative arts therapy modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Participate patients need to be (a) diagnosed with a disorder that requires an allogeneic stem cell transplant, (b) scheduled for allogeneic stem cell transplant and expected to be admitted for ~3-4 weeks
2. Aged 18 years or older
3. Score ≥1 on the distress thermometer
4. Have access to a smartphone, tablet, or computer with internet capability in order to complete study surveys via Microsoft Forms and to connect to a music streaming platform via website or app
5. Able to provide informed consent.

Exclusion Criteria:

1. Individuals with significant and active cognitive (e.g., major cognitive impairment), psychiatric (e.g., active psychosis), or medical conditions (e.g., untreated significant hearing impairments) that would prevent the ability to provide informed consent or participate in the music listening intervention
2. Individuals without access to music streaming via smartphone, tablet, or computer and have access to internet.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM): Mindful Music Listening Group mean >=4 at follow-up | Post-intervention follow-up at 4 weeks post inpatient admission
  Feasibility of Intervention Measure (FIM): The FIM has 4 items ranging from 1 (Completely Disagree) to 5 (Completely Agree). Higher scores indicate greater feasibility. Mindful Music Listening (MML) group mean score >=4 (reflective of an average response of "Agree") at post-intervention will be considered the benchmark for determining that the intervention was feasible, acceptable, and/or appropriate.
Acceptability of Intervention Measure (AIM): Mindful Music Listening Group mean >=4 at follow-up | Post-intervention follow-up at 4 weeks post inpatient admission
  Acceptability of Implementation Measure (AIM): The Implementation Appropriateness Measure (IAM) (Weiner et al., 2017) Higher scores indicate greater appropriateness. Mindful Music Listening (MML) group mean score >=4 (reflective of an average response of "Agree") at post-intervention will be considered the benchmark for determining that the intervention was feasible, acceptable, and/or appropriate.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) | Post-intervention follow-up at 4 weeks post inpatient admission
  To measure physical, emotional, functional, and social well-being the Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT (Version 4)) will be used. The study team chose the FACT-BMT because it contains FACT-G (a cancer specific health-related quality of life measure) and additional BMT-specific items. It contains a total of 47 items that are separated into the following domains and scored on a Likert scale: physical well-being, social and family well-being, relationship with doctor, emotional well-being, functional well-being, and additional concerns. This measure is used on patients receiving an autologous or allogeneic HSCT to treat a hematological condition.
Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale (HADS-A total score) and Depression Subscale (HADS-D total score) | Post-intervention follow-up at 4 weeks post inpatient admission
  The Hospital Anxiety and Depression Scale (HADS) is a validated means of measuring symptoms of depression and anxiety. It consists of 14 items (7 items for each subscale) on a 4-point Likert scale (ranging from 0-3). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). After adjusting for six items that are reversed scored, all responses are summed to obtain the two subscales. A cut-off score of 8 is utilized (Bjelland, Dahl, Haug, & Neckelmann, 2002). The scale was chosen because it does not include somatic aspects of depression (e.g., insomnia and weight loss) which are often present in patients diagnosed with blood cancers, rather the scale is focused on anhedonia. Overall, it has demonstrated satisfactory psychometric properties in various groups including cancer inpatients (Annunziata, Muzzatti, & Altoè, 2011).
Five Facet Mindfulness Questionnaire- 15 item short form (FFMQ-15) | Post-intervention follow-up at 4 weeks post inpatient admission
  The Five Facet Mindfulness Questionnaire (FFMQ-15) is a short form (15 items) of the 39-item FFMQ (Baer et al., 2006). It includes the same five facets as the long form: Observing, Describing, Acting with Awareness, Non-Judging of inner experience, and Non-Reactivity to inner experience. The 15 question self-report scale measures mindfulness with regards to thoughts, experiences, and actions in daily life (Baer, Carmody, & Hunsinger, 2012). The questions are scored on a 1-5 Likert scale from "never or very rarely true" to "very often or always true." Higher scores are indicative of someone who is more mindful in their everyday life. The factor structure and psychometric properties of the FFMQ-15 were tested by Gu et al. (2016). This questionnaire will be used to illustrate whether participants that are more mindful in their everyday lives respond more to a music listening intervention and whether the intervention impacts their ability to be mindful.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Olex, Psy.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No